CLINICAL TRIAL: NCT05887427
Title: Acute Effect of Neural Mobilization in Cervical Radiculopathy: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Büşra Sökmen Yıldırım, physiotherapist, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Üsküdar Üniversitesi
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Cervical Radiculopathy
Keywords: NEURAL MOBİLİSATİON,CERVİCAL RADİCULOPATHY,
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilisation Group (NMG) (Experimental): The neural mobilisation group received one session of conservative physiotherapy and neural mobilization at the end of the session. The content of the conservative program was the same in both groups. Before the neural mobilization application, a nerve stretching test was performed to provide a specific stretching position for each nerve and the patient was asked if he/she had any complaints. After adjusting the intensity of the neural mobilization tension, all participants were asked if they felt numbness, tension or tingling sensation in the nerve. When the symptoms were at a level that did not bother the patient, the nerve was held in that position for 10 seconds and then the nerve was left in the relaxation position. Each neural mobilization was performed in 10 repetitions.
  Interventions: Other: Neural Mobilisation
- Control Group (CG) (Active Comparator): Control group patients received one session of conservative physiotherapy program. The conservative program consisted of 20 minutes of heat application to the cervical region, 20 minutes of Transcutaneous Electrical Stimulation (TENS) application and 5 minutes of ultrasound application.
  Interventions: Other: Conservative physiotherapy

INTERVENTIONS:
Other: Neural Mobilisation — Transcutaneous Electrical Stimulation, hotpack, ultrasound and neural mobilization(radial,ulnar,median)
  Arms: Neural Mobilisation Group (NMG)
Other: Conservative physiotherapy — Hotpack,Transcutaneous Electrical Stimulation ,Ultrasound
  Arms: Control Group (CG)

SUMMARY:
The aim of this study was to investigate the immediate effect of neural mobilization techniques, one of the manual therapy methods that can be used in the treatment of cervical radiculopathy.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled experimental study and was conducted in the Physiotherapy and Rehabilitation Department of Istanbul Medicana International Hospital. Population: The study included patients diagnosed with cervical disc herniation who were referred to physiotherapy sessions by a physician Patients were assigned to the Control Group(CG) or Neural Mobilization Group(NMG) by simple randomization. The control group received conventional physiotherapy while the neural mobilization group received neural mobilization of the ulnar median and radial nerves. The pain of the patients was evaluated with Numeric Pain Rating Sacale (NPRS) and Neuropathic Pain Questionnaire (NPQ) at the beginning and end of the intervention, while hand grip strength and pinch grip strength were evaluated with digital hand dynamometer (JAMAR Plus Digital Hand Dynamometer) and digital pinchmeter (JAMAR Plus Pinch Gauge). Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting the following criteria were included in the study: age between 18 and 65 years, referred to physiotherapy with a diagnosis of cervical disc herniation, self-reported neck pain with a visual analog scale (VAS) score of more than 5, presence of pain radiating from the neck to the arm, and at least 3 of the following tests were positive: Spurling's Test, Upper Extremity Tension Test-1, Distraction Test, and ipsilateral cervical rotation less than 60 degrees. These tests were assessed by a trained examiner according to standardized procedures

Exclusion Criteria:

* Exclusion criteria were surgical intervention in the head and neck region, history of fracture in the head and neck region, known chronic disease, infection and structural disorders in the bone and soft tissue in the cervical spine, malignancy and severe osteoporosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 2 Month
  Pain in the neck region of the participants was evaluated using NPRS before and after the intervention. On this scale, patients were asked to mark the pain they felt on a 10 cm scale. Accordingly, the participants marked the range of values "0" was no pain, and "10" was the most severe.
Neuropathic Pain Questionnaire (NPQ) | 2 Month
  Before and after the intervention, the characteristics and severity of the patients' pain were evaluated with the Neuropathic Pain Questionnaire. This scale was used for initial screening of patients with pain. It has the ability to provide a quantitative measurement for the symptoms that are important in the diagnosis and evaluation of neuropathic pain. In the questionnaire consisting of 12 questions, 10 questions were asked about the nature of pain and the other two questions about changes in sensitivity.

SECONDARY OUTCOMES:
Hand Grip Strength | 2 Month
  A digital hand dynamometer (JAMAR Plus Digital Hand Dynamometer) , was used to measure hand grip strength.. The test was performed in an upright sitting position, 3 measurements were performed with one-minute intervals between each measurement and the averages were recorded. For painless grip strength, patients were asked to squeeze the dynamometer until they felt discomfort before and after treatment.The shoulder was in adduction and neutral position, elbow in 90° flexion, forearm in neutral position and wrist in 0 -30° extension and 0-15° ulnar deviation position while the patients were sitting in a chair with their arms supported.Both hands were measured separately.
Pinch Grip Strength | 2 Month
  Pinch grip (two-point grip) strength was evaluated with a pinch meter (JAMAR Plus Pinch Gauge). The application was performed comparatively in both extremities; patients were sitting in a chair with support, shoulder in adduction and neutral position, elbow in 90˚ flexion, forearm in neutral position, wrist in 0-30˚ extension and 0-15˚ ulnar deviation position.Measurements were taken before and after the intervention. Three measurements were made with one minute intervals between each measurement and the averages were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: BERNA KARAMANCIOĞLU, Study Director — berna.karamancioğlu@uskudar.edu.tr
Locations (1):
- Üsküdar University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No